CLINICAL TRIAL: NCT02117141
Title: A Pilot Study in Healthy Volunteers to Assess the Rate and Extent of Absorption of Hydrocodone From 20 mg Hydrocodone Bitartrate Extended-Release (HC-ER) Capsules, in Both Fed and Fasted States
Brief Title: To Assess the Rate and Extent of Absorption of Hydrocodone From 20 mg Hydrocodone Bitartrate Extended-Release Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ELN-0302002
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Food Effect; Pharmacokinetics
MeSH Terms: interventions — Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HC-ER 20 mg capsule (fasted) (Experimental): Single oral dose of a HC-ER 20 mg capsule (fasted)
  Interventions: Drug: HC-ER 20 mg capsule (fasted)
- HC-ER 20 mg capsule (fed) (Experimental): Single oral dose of HC-ER 20mg capsule (fed)
  Interventions: Drug: HC-ER 20 mg capsule (fed)

INTERVENTIONS:
Drug: HC-ER 20 mg capsule (fasted) — Single oral dose HC-ER 20 mg capsule after overnight fast (fasted)
  Other Names: Zohydro ER
  Arms: HC-ER 20 mg capsule (fasted)
Drug: HC-ER 20 mg capsule (fed) — Single oral dose HC-ER 20 mg capsule after high fat meal (fed)
  Other Names: Zohydro ER
  Arms: HC-ER 20 mg capsule (fed)

SUMMARY:
* Assess the rate and extent of absorption of hydrocodone from a 20 mg HC-ER capsule in both fed and fasted states
* Evaluate the safety and tolerability of the test compound administered orally

DETAILED DESCRIPTION:
Safety parameters assessed included medical history, physical examination, vital signs, 12-lead ECGs, clinical laboratory testing and adverse event assessment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers.
* Aged greater than 18 and less than 45 years.
* Were medically healthy with no clinically significant abnormality on the basis of medical history, physical examination and laboratory evaluations
* Volunteer consented to participate in the study.
* Female volunteers were included if they were surgically sterile, or using an acceptable method of birth control defined as either oral, injectable, implantable, or barrier methods of contraception (ie, diaphragm with spermicidal cream, intrauterine device (IUD) with spermicidal cream or condom with spermicidal cream).

Exclusion Criteria:

* Participants were in a clinical trial within the previous 90 days or participants in a narcotic analgesic study within the previous 12 months.
* Deviation in excess of 10% from the ideal body weight for height according to the Metropolitan Life Insurance Tables (1983 edition).
* History of drug or alcohol abuse at any time in the past
* History of hypersensitivity to the study drug or similar compounds or to acetaminophen.
* Therapeutic use (for any reason) of narcotic analgesics within the previous year.
* Subjects who used tricyclic antidepressants or monoamine oxidase inhibitors at any time in the past.
* Subjects with a history of, or clinical signs suggestive of, chronic obstructive airways disease.
* Receipt of any prescription medication (except birth control) within 2 weeks prior to entry into the study or receipt of non-prescription or over-the-counter medication within one week of study commencement. (Vitamin supplements were acceptable).
* Blood donation within the 90 days previous to study entry.
* Female volunteers with a positive serum pregnancy test, or at risk of becoming pregnant during the study.
* Volunteers with a history of smoking (must not have smoked within the last 6 months).
* Volunteers with any clinical/biochemical impairment of liver function, or receipt of known hepatic enzyme inducing or inhibiting agents within 30 days prior to entry into the study.
* History or presence of significant hepatic, renal, endocrine, cardiac, nervous, gastrointestinal, pulmonary or metabolic disorders.
* Any condition or history that the investigator considered might increase the risk to the volunteer or interfere with the evaluation of data.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2002-06; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Assess the rate and extent of absorption of hydrocodone from a 20 mg HC-ER capsule in both fed and fast states | Day 1-2

CONTACTS AND LOCATIONS:
Overall Officials: A. Johnston Stewart, MB, MRCGP, Principal Investigator — Zogenix, Inc.